CLINICAL TRIAL: NCT06786676
Title: A Randomized, Double-blind, Placebo-controlled, Single- and Multiple-oral Administration, Phase 1 Clinical Trial to Investigate the Safety, Tolerability, and Pharmacokinetics of AS-S603 in Healthy Korean or Caucasian Adults and Korean Elderly People
Brief Title: A Phase 1 Clinical Trial to Investigate the Safety, Tolerability, and Pharmacokinetics of AS-S603 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Amyloid Solution Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AS-S603-P101
Record Dates: First submitted 2025-01-08; First posted 2025-01-22 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: AD; Alzheimer Disease; AS-S603; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (AS-S603) (Experimental): Korean and Caucasian Participants
  Interventions: Drug: AS-S603
- Placebo group (Placebo of AS-S603) (Placebo Comparator): Korean and Caucasian Participants
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AS-S603 — Oral administration of AS-S603 tablet
  Arms: Test group (AS-S603)
Drug: Placebo — Oral administration of Placebo tablet
  Arms: Placebo group (Placebo of AS-S603)

SUMMARY:
This trial is a randomized, double-blind, placebo-controlled, single- and multiple-oral administration, phase 1 clinical trial to investigate the safety, tolerability, and pharmacokinetics of AS-S603 in healthy Korean or Caucasian adults and Korean elderly people.

AS-S603 is an orally administered agent developed by Amyloid Solution Inc to treat Alzheimer's disease (AD). It is a small molecule compound that targets and dissolves amyloid-beta (Aβ) and tau aggregates, two key pathologies present in the extracellular and intracellular spaces of brain cells in AD.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Korean adult volunteers aged 19 to 50 years at the time of screening (single dose study)
* Healthy Korean or Caucasian adult volunteers aged 19 to 50 years at the time of screening (multiple dose study dose groups 1-4)
* Healthy elderly Korean volunteers aged 65 to 85 years at the time of screening (multiple dose study dose group 5)
* Individuals with a body weight of ≥ 50.0 kg and ≤ 90.0 kg and a body mass index of ≥ 18.5 kg/m2 and ≤ 29.9 kg/m2 at the time of screening
* Individuals who have given written consent on a voluntary decision to participate and agree to adhere to the precautions after being fully informed of and completely understanding this clinical trial

Exclusion Criteria:

* Individuals with a clinically significant disease or history in hepatobiliary, renal, nervous, immune, respiratory, endocrine, hemato-oncology, cardiovascular, urinary system, or psychiatric disorder.
* Individuals with a history of a gastrointestinal disorder or surgery that may affect the safety, pharmacokinetic and pharmacodynamic evaluation of the investigational product
* Individuals who answered 'yes' to any question on the Columbia Suicide Severity Rating Scale administered at the time of screening
* Individuals with hypersensitivity or a history of clinically significant hypersensitivity to AS-S603 and the same class or other drugs (aspirin, antibiotics, etc.)
* Individuals with a positive result in the serology test (hepatitis B, hepatitis C, human immunodeficiency virus test, syphilis test)
* Individuals with a history of drug abuse or a positive urine screening for any drug of concern for abuse
* Individuals who exhibited the following results on vital signs measured at a sitting position after resting, during the screening tests: Systolic blood pressure < 80 mmHg or ≥ 140 mmHg, Diastolic blood pressure < 45 mmHg or ≥ 90 mmHg
* Individuals who exhibited QTcB interval > 450 msec (male), 470 msec (female), or clinically significant abnormal findings in rhythm on an electrocardiogram during the screening tests
* Individuals who exhibited any of the following results on the clinical laboratory test during the screening tests, including additional tests: Aspartate transaminase or alanine transaminase > 60 IU/L, Estimated glomerular filtration rate < 90 mL/min/1.73m2
* Individuals who had taken any prescription drug or herbal medicine within 2 weeks, or any Over-The-Counter (OTC) drugs, dietary supplements including liver supplements, or vitamin supplements within 1 week prior to the scheduled first administration of investigational product, or are expected to take them
* Individuals who had taken an inducer or inhibitor of any drug metabolic enzyme, such as barbiturates or clarithromycin, within 1 month prior to the scheduled first administration of investigational product
* Individuals who have participated and administered investigational product in another clinical trial within 6 months prior to the scheduled first administration of investigational product
* Individuals who donated whole blood within 2 months, donated blood components within 1 month, or received a blood transfusion within 1 month prior to the scheduled first administration of investigational product
* Current smokers
* Individuals who engage in persistent alcohol consumption or are not able to avoid alcohol consumption from 3 days prior to the scheduled first administration of investigational product until the end of the clinical trial.
* Individuals who have consumed excessive caffeine or are not able to avoid consuming caffeine-containing foods from 3 days prior to the scheduled first administration of investigational product until the end of the clinical trial.
* Individuals who have consumed grapefruit, grapefruit juice, or grapefruit-containing foods or cannot avoid consuming grapefruit-containing foods from 3 days prior to the scheduled first administration of investigational product until the end of the clinical trial.
* Individuals with unusual dietary habits or who cannot adhere to the standardized diet provided by the institution during the confinement period.
* Women of childbearing potential, individuals whose menstrual period was not confirmed at screening, with a positive urine pregnancy test, or who do not agree to a highly effective contraceptive method for at least 30 days after the last investigational product administration.
* Men who do not agree to use condoms and ensure that their female partners use a highly effective contraceptive method throughout the entire clinical trial period and for at least 90 days after the last administration of investigational product.
* Individuals who do not agree to refrain from donating sperm or egg throughout the entire clinical trial period and for at least 90 days after the last administration of investigational product.
* Individuals who cannot undergo cerebrospinal fluid (CSF) tapping (for groups requiring CSF tapping)
* Individuals determined to be ineligible for participation in the clinical trial by the investigators due to other reasons

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 88 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events (AEs) | Up to Day 27
Maximum observed concentration (Cmax) | Up to Day 18
Time of maximum observed concentration (Tmax) | Up to Day 18
Terminal half-life (t1/2) | Up to Day 18
Area under the concentration-time curve from the time of dosing to the time of the last measurable concentration (AUClast) | Up to Day 18
Area under the concentration-time curve from the time of dosing extrapolated to infinity (AUCinf) | Up to Day 18

OTHER OUTCOMES:
pTau217 concentration and Aβ42/40 ratio in plasma and cerebrospinal fluid (CSF) | Up to day 27
  Exploratory pharmacodynamic evaluation based on pTau217 concentration and Aβ42/40 ratio in plasma and CSF

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital Clinical Trial Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No